CLINICAL TRIAL: NCT01863186
Title: Phase 3, Randomized, Multicenter, Double-Blind, Placebo-Controlled, Efficacy, Safety, and Dose-Response Study of Lofexidine for Treatment of Opioid Withdrawal (Days 1-7) Followed by Open-Label, Variable Dose Lofexidine Treatment (Days 8-14)
Brief Title: Efficacy, Safety and Dose-Response Study Followed by Open-Label Study of Lofexidine Treatment of Opioid Withdrawal
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: USWM, LLC (dba US WorldMeds) (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: USWM-LX1-3003-1; 1U01DA033276-01A1 (NIH)
Record Dates: First submitted 2013-05-22; First posted 2013-05-27 (Estimated); Results first posted 2021-02-04 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-02

CONDITIONS: Opioid Dependence; Acute Opioid Withdrawal Syndrome
Keywords: lofexidine; opioid dependence; acute withdrawal syndrome; opioid withdrawal
MeSH Terms: conditions — Opioid-Related Disorders | interventions — lofexidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Lofexidine HCl (2.4mg dose) (Active Comparator): 225 subjects will be randomized to receive 2.4 mg total daily dose of lofexidine HCl during the double-blind period of the study. Subjects will take 4 tablets QID for a total daily dose of 2.4 mg (one tablet in each dose will be a placebo tablet to maintain the blind) for up to 7 days.
  Interventions: Drug: Lofexidine HCl; Drug: Placebo
- Lofexidine HCl (3.2mg dose) (Active Comparator): 225 subjects will be randomized to receive 3.2 mg total daily dose of lofexidine HCl during the double-blind period of the study. Subjects will take 4 tablets QID for a total daily dose of 3.2 mg for up to 7 days.
  Interventions: Drug: Lofexidine HCl
- Placebo (Placebo Comparator): 150 subjects will be randomized to receive placebo during the double-blind period of the study. Subjects will take 4 tablets QID for up to 7 days.
  Interventions: Drug: Placebo
- Open Label Lofexidine HCl (Other): During the open-label portion of the study, subjects will be given the option to receive lofexidine HCl tablets for up to 7 days. Dosing regimens are at the discretion of the Investigator.
  Interventions: Drug: Open Label Lofexidine HCL

INTERVENTIONS:
Drug: Lofexidine HCl — Lofexidine HCl tablets will be available in 0.2 mg tablets. Lofexidine will be provided in total daily doses as indicated during the double blind portion of the study.
  Arms: Lofexidine HCl (2.4mg dose); Lofexidine HCl (3.2mg dose)
Drug: Placebo — Lofexidine-matching tablets without the active pharmaceutical ingredient will be provided as 4 tablets QID during the double-blind portion of the study to subjects randomized to placebo.
  Arms: Lofexidine HCl (2.4mg dose); Placebo
Drug: Open Label Lofexidine HCL — Lofexidine HCl tablets will are available in 0.2 mg tablets. During the optional open-label portion of the study, Lofexidine HCl can be prescribed at the discretion of the Investigator but total daily dose will not exceed 3.2 mg.
  Arms: Open Label Lofexidine HCl

SUMMARY:
The purpose of this study is to look at the efficacy and safety for lofexidine hydrochloride, an alpha-2 adrenergic agonist under development for the treatment of acute withdrawal from short-acting opioids. The study takes place in 2 parts: a 7-day inpatient double-blind treatment portion where subjects will be randomly assigned to one of three doses of study medication (2.4 mg total daily dose of lofexidine, 3.2 mg total daily dose of lofexidine, or placebo) followed by an optional open-label treatment period where subjects will be inpatient or outpatient and receive lofexidine at variable dosing for up to an additional 7 days. The Investigator hypothesizes that subjects will achieve maximum treatment effect with tolerable side effects at the 3.2 mg total daily dose and that both the 3.2 mg and 2.4 total daily doses will show better efficacy over placebo in treating symptoms of acute opioid withdrawal.

DETAILED DESCRIPTION:
This is a Phase 3, two-part, multicenter study to evaluate the dose-response, efficacy, and safety of lofexidine in alleviation of symptoms in subjects undergoing total and abrupt withdrawal from short-acting opioids. Any subject dependent on short-acting opioids (the primary projected indication for lofexidine) about to undergo opioid withdrawal will be eligible. Subjects will be evaluated for their compliance with protocol inclusion/exclusion criteria during a screening period, lasting up to 7 days.

The first part of the study will use an inpatient, randomized, double-blind, and placebo-controlled design (Days 1-7) followed by a second part, an open-label continuation treatment (Days 8-14). A total of 600 subjects will be randomized to receive lofexidine 2.4 mg total daily dose (0.6 mg QID), lofexidine 3.2 mg total daily dose (0.8 mg QID), or matching placebo in a 3:3:2 ratio (225:225:150) for 7 days (i.e., during the most intense stage of withdrawal). During the second part of the study (Days 8-14), all subjects, regardless of their treatment assignment (which will remain double-blinded), who successfully meet the definition for "completer" based on Days 1-7 (i.e., receives at least one dose of study medication on Day 7 and completes the 3.5-hour post-dose SOWS-Gossop assessment on Day 7), will be eligible to receive open-label, variable dose lofexidine treatment (as determined by the Site Investigator, but not to exceed 3.2 mg/day) for up to an additional 7 days in either an inpatient or outpatient setting depending on the wishes of the investigator and the subject. No subject will receive lofexidine for more than 14 days total from the onset of abstinence. There will be no initial dose run-up and no mandated terminal dose taper.

Efficacy and safety assessments will be made daily throughout the study. Safety will be assessed by evaluation of adverse event, clinical labs, electrocardiograms (with special attention to QTc), vital signs, physical exam data, and the Columbia-Suicide Severity Rating Scale. Efficacy will be evaluated daily by subject- and observer-completed scales including the Short Opiate Withdrawal Scale of Gossop (SOWS-G)(the primary outcome measure is SOWS-G score area under the curve for Days 1-7), the Clinical Opiate Withdrawal Scales (COWS), Objective Opiate Withdrawal Scale (OOWS-Handelsman), the Visual Analog Scale for Efficacy (VAS-E), and the Modified Clinical Global Impressions scales for efficacy and side effects. Efficacy will also be evaluated by study retention, completion rates, concomitant medication use, incidence of withdrawal-related Adverse Events (AEs), and subject treatment status 30 days post last dose of study medication. Qualitative urine drug screening will be done every other day to monitor for contraband (inpatient setting) or illicit (outpatient setting) drug use. Upon a subject's exit from the study, Study Discontinuation/End of Study assessments will be done.

During the study, study drug compliance will be documented in the source daily. During the first part of the study (Days 1-7), subjects will be inpatient and each dose of study medication will be administered by study site personnel and recorded in the source. Study medication will be dosed QID at 8 AM, 1 PM, 6 PM and 11 PM. During the second part of the study (Days 8-14), subjects who remain inpatient will be administered each dose of study medication by study site personnel and dosing will be captured in the source. Subjects who complete the second part of the study on an outpatient basis will return to the clinic daily for study assessments. During the open-label period, subjects will be dispensed 1-2 days worth of study drug, as needed to allow for flexibility in scheduling daily visits, to get them through until they are supposed to return the following day for additional study assessments and dosing.

Study medication will be held if vital signs meet any of the following criteria: Resting (sitting or recumbent, if required, for treatment of an adverse event): Systolic blood pressure <90 mmHg and >20% below screen value; Diastolic blood pressure <50 mmHg and >20% below screen value; Heart rate <50 bpm and >20% below screen value; and Symptoms of hypotension and/or bradycardia (e.g., lightheadedness, dizziness, syncope).Orthostatic (after standing for 3 minutes): Systolic blood pressure diastolic blood pressure, or pulse >25% below recumbent values.

A subject will be discontinued from the study if any of the following criteria are met: Systolic blood pressure <70 mmHg and >20% below screen value; Diastolic blood pressure <40 mmHg and >20% below screen value; Heart rate <40 bpm and >20% below screen value; QTc >500 msec or >25% above screen value for both males and females; Syncope; Subject misses more than 2 doses in 24 hours during Days 1-7 prior to meeting "completer" criteria (i.e., receives at least one dose of study medication on Day 7 and completed the 3.5-hour post-dose SOWS-Gossop assessments on Day 7); Subject misses a total of 6 doses during Days 1-7 prior to meeting "completer" criteria (i.e., receives at least one dose of study medication on Day 7 and completed the 3.5-hour post-dose SOWS-Gossop assessments on Day 7); Concomitant medication use (other than alumina, magnesia, and simethicone) for intolerable nausea and emesis.

Subjects should be discontinued from the study for any of the reasons listed below, and the event should be recorded as an Adverse Event (AE) and the subject followed until medically stabilized to the satisfaction of the attending physician: New onset of clinically significant abnormal ECG (e.g., second or third degree heart block or uncontrolled arrhythmia, prolonged QTcF interval); Persistent symptomatic hypotension (e.g., hypotension not responding to bed rest or fluids); Single occurrence of symptomatic bradycardia (as assessed by the Investigator, regardless of blood pressure) associated with chest pain, shortness of breath, or decreased level of consciousness; Persistent hypertension - blood pressure ≥185/110 mmHg recorded on 3 separate occasions taken at least 5 minutes apart AND within a 1-hour time period. If all 3 readings are ≥185/110 mmHg (either systolic ≥185 mmHg or diastolic ≥110 mmHg) the subject must be terminated; Medical Intervention for Cardiovascular Event: Any medical intervention (nonmedication or medication inclusive) used for the treatment of any cardiovascular event, with the exception of a positional intervention in subjects displaying hypotension; Any other clinically significant cardiovascular signs or symptoms that would place the subject at risk.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age.
* Currently dependence, according to the Mini International Neuropsychiatric Interview (M.I.N.I.) [17, 18], on any opioid with a half-life similar to heroin or morphine, including Vicodin®, Lortab®, Lorcet®, Percocet®, Percodan®, Tylox®, or Hydrocodone (by any route of administration), or oxycodone (oxycodone and oxycodone time-released formulation when crushed and snorted, injected or swallowed after chewing).
* Seeking treatment for opioid dependence.
* Score of ≥2 on the Objective Opiate Withdrawal Scale (OOWS-Handelsman) at Baseline.
* Reported use of heroin, morphine, or any opioid with a half-life similar to heroin or morphine for at least 21 of the past 30 days.
* Urine toxicology screen positive for opioids but negative for methadone and buprenorphine.
* Females of childbearing potential must agree to using birth control methods and must have had documented proof.
* Able to verbalize understanding of the consent form, able to provide written informed consent, verbalize willingness to complete study procedures, and pass the study consent quiz with 100% accuracy (if necessary, quiz may be administered more than one time).

Exclusion Criteria:

* Female subject who is pregnant or lactating.
* Self-reported use of methadone or buprenorphine in the past 14 days.
* Serious medical illnesses including, but not limited to: seizures, pancreatic disease, liver disease, exposure to a hepatitis virus, and positive hepatitis results.
* Psychiatric disorder, based on the M.I.N.I., including but not limited to dementia or any disorder that, in the opinion of the study physician requires ongoing treatment that would make study participation unsafe or which would make treatment compliance difficult.
* Self-reported acquired immune deficiency syndrome (AIDS) or self-reported human immunodeficiency virus (HIV) positive status and taking retroviral medications currently or within the past 4 weeks.
* Abnormal cardiovascular exam at screening and before randomization, including any of the following: clinically significant abnormal electrocardiogram (ECG) (e.g., second or third degree heart block, uncontrolled arrhythmia, or QTcF interval greater than 450 msec for males and greater than 470 msec for females); heart rate less than 55 bpm or symptomatic bradycardia; systolic blood pressure (SBP) less than 95 mmHg or symptomatic hypotension; diastolic blood pressure (DBP) less than 65 mmHg; blood pressure (BP) greater than 155/95 mmHg; and prior history of myocardial infarction.
* Clinically significant abnormal laboratory values.
* Requiring any of the following medications currently or within the past 4 weeks: psychotropics (including sedatives/hypnotics, antidepressants, neuroleptics), prescription analgesics (excluding those listed in inclusion criterion #2 above), anticonvulsants, antihypertensives, antiarrhythmics, antiretroviral, and cholesterol lowering medications. Nicotine replacement therapy (patch, inhaler, gum, or nasal spray) will be allowed for nicotine-dependent subjects. Note: Use of a short-acting benzodiazepine (e.g., oxazepam) for insomnia during Days 8 14 will not disqualify a subject.
* Currently dependent (based on the M.I.N.I.) on any psychoactive substance (other than that listed in inclusion criterion #2, caffeine or nicotine) that requires detoxification.
* Donated blood within the last 8 weeks.
* Participated in an investigational drug study within the past 3 months.
* Has "poor" veins that even a single venipuncture cannot be obtained during screening.
* Active tuberculosis (positive tuberculin test and/or confirmatory diagnostic chest x-ray).
* Active syphilis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 603 (Actual)
Dates: Start 2013-06; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles W Gorodetzky, MD, PhD, Principal Investigator — US WorldMeds
Locations (18):
- United States (18):
  - Clovis, California
  - Escondido, California
  - San Diego, California
  - Miami, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Oak Park, Illinois
  - Lake Charles, Louisiana
  - Baltimore, Maryland
  - Flowood, Mississippi
  - St Louis, Missouri
  - Dayton, Ohio
  - Mason, Ohio
  - Austin, Texas
  - Dallas, Texas
  - DeSoto, Texas
  - Orem, Utah
  - Salt Lake City, Utah

REFERENCES:
- [Derived] Alam D, Tirado C, Pirner M, Clinch T. Efficacy of lofexidine for mitigating opioid withdrawal symptoms: results from two randomized, placebo-controlled trials. J Drug Assess. 2020 Jan 8;9(1):13-19. doi: 10.1080/21556660.2019.1704416. eCollection 2020. PMID 32002194
- [Derived] Darpo B, Pirner M, Longstreth J, Ferber G. Effect of lofexidine on cardiac repolarization during treatment of opioid withdrawal. Drug Alcohol Depend. 2019 Dec 1;205:107596. doi: 10.1016/j.drugalcdep.2019.107596. Epub 2019 Sep 27. PMID 31606589
- [Derived] Fishman M, Tirado C, Alam D, Gullo K, Clinch T, Gorodetzky CW; CLEEN-SLATE Team. Safety and Efficacy of Lofexidine for Medically Managed Opioid Withdrawal: A Randomized Controlled Clinical Trial. J Addict Med. 2019 May/Jun;13(3):169-176. doi: 10.1097/ADM.0000000000000474. PMID 30531234

RESULTS

PARTICIPANT FLOW:
Groups:
- DB: Lofexidine HCl 2.4mg Dose: Participants were randomized to receive 2.4 mg total daily dose of lofexidine HCl during the double-blind period of the study. Subjects will take 4 tablets QID for a total daily dose of 2.4 mg (one tablet in each dose will be a placebo tablet to maintain the blind) for up to 7 days.
- DB: Lofexidine HCl 3.2mg Dose: Participants were randomized to receive 3.2 mg total daily dose of lofexidine HCl during the double-blind period of the study. Subjects will take 4 tablets QID for a total daily dose of 3.2 mg for up to 7 days.
- DB: Placebo: Participants were randomized to receive placebo during the double-blind period of the study. Subjects will take 4 tablets QID for up to 7 days.
  Placebo: Lofexidine-matching tablets without the active pharmaceutical ingredient will be provided as 4 tablets QID during the double-blind portion of the study to subjects randomized to placebo.
- OL: All Lofexidine HCl: Participants were given the option to receive lofexidine HCl tablets for up to 7 additional days, following the double blind period. Dosing regimens are at the discretion of the Investigator, but total daily dose will not exceed 3.2 mg.
Period: Double-blind Phase
Arm/Group | DB: Lofexidine HCl 2.4mg Dose | DB: Lofexidine HCl 3.2mg Dose | DB: Placebo | OL: All Lofexidine HCl
Started | 229 (Original number of 230. One participant was randomly assigned into the study, but not dosed.) | 222 | 151 | 0
Completed | 95 | 88 | 42 | 0
Not Completed | 134 | 134 | 109 | 0
Period: Open-label Phase
Arm/Group | DB: Lofexidine HCl 2.4mg Dose | DB: Lofexidine HCl 3.2mg Dose | DB: Placebo | OL: All Lofexidine HCl
Started | 0 | 0 | 0 (No placebo group in the Open-label Phase.) | 83 (36 from 2.4 mg group, 28 from 3.2mg group, and 19 from Placebo continued to the Open-label phase.)
Completed | 0 | 0 | 0 | 70
Not Completed | 0 | 0 | 0 | 13

BASELINE CHARACTERISTICS:
Population: Demographic Characteristics of modified intent-to-treat "mITT" Population (excludes one subject who randomized but never received study drug)
Groups:
- Total: Total of all reporting groups
Arm/Group | DB: Lofexidine HCl 2.4mg Dose | DB: Lofexidine HCl 3.2mg Dose | DB: Placebo | Total
Number analyzed (Participants) | 229 | 222 | 151 | 602
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (10.8) | 35 (10.5) | 36 (11.9) | 35 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 64 | 44 | 175
  Male | 162 | 158 | 107 | 427
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 28 | 22 | 83
  Not Hispanic or Latino | 196 | 194 | 129 | 519
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2 | 4
  Asian | 1 | 3 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 3 | 5
  Black or African American | 54 | 48 | 26 | 128
  White | 169 | 158 | 117 | 444
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 9 | 2 | 16
Body weight [Mean (Standard Deviation); unit: kg] | 76.0 (16.88) | 76.1 (16.59) | 76.0 (14.94) | 76.1 (16.29)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 25.1 (4.71) | 25.1 (5.32) | 25.1 (4.63) | 25.1 (4.92)

OUTCOME MEASURES:

1. Primary Outcome: Difference Between the Overall Means From Short Opiate Withdrawal Scale of Gossop (SOWS-Gossop) Scores
Description: The SOWS-Gossop was completed by the mITT population subject at baseline, once daily at 3.5 hours after the first dose of the study medication on Days 1 to 7. It consists of 10 items that are scored on a 4-point scale; 0=none, 1=mild, 2=moderate, and 3=severe. The overall score is the simple sum of the 10-item scores (minimum overall score of 0, maximum score of 30). Higher individual scores on the scale indicate greater symptom severity. However, as the outcome measure is a difference from placebo, a lower number indicates a better outcome.
  mITT population: all randomized subjects who received at least 1 dose of study medication
Time Frame: Days 1 through 7
Population: mITT population Participants Analyzed does not match the Participant Flow because of missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DB: Lofexidine HCl 2.4mg Dose | DB: Lofexidine HCl 3.2mg Dose | DB: Placebo
Number analyzed (Participants) | 229 | 222 | 151
score on a scale
  Day 1: number analyzed (Participants) | 227 | 220 | 148
  Day 1 | 7.8 (6.00) | 7.6 (6.75) | 9.4 (6.81)
  Day 2: number analyzed (Participants) | 191 | 183 | 106
  Day 2 | 10.2 (6.83) | 9.9 (7.38) | 13.9 (8.29)
  Day 3: number analyzed (Participants) | 154 | 139 | 73
  Day 3 | 7.6 (5.53) | 7.4 (6.34) | 10.9 (6.76)
  Day 4: number analyzed (Participants) | 128 | 121 | 62
  Day 4 | 5.7 (5.32) | 5.5 (5.36) | 9.2 (6.81)
  Day 5: number analyzed (Participants) | 110 | 112 | 53
  Day 5 | 4.7 (4.60) | 4.5 (4.96) | 6.4 (5.91)
  Day 6: number analyzed (Participants) | 100 | 96 | 47
  Day 6 | 3.6 (3.97) | 3.2 (4.10) | 4.4 (5.80)
  Day 7: number analyzed (Participants) | 101 | 96 | 44
  Day 7 | 2.7 (3.45) | 2.3 (3.23) | 2.7 (4.60)
Statistical Analysis 1: Comparison: DB: Lofexidine HCl 2.4mg Dose vs DB: Placebo; Due to the amount of missing data a pattern mixture model (or Jump to Reference) was utilized. The SOWS-Gossop total scores were log transformed. Each subjects available data Days 1-7 were included. The datasets created by the pattern mixture model were analyzed using a Mixed Model Repeated Measures model that included fixed effects for treatment group, baseline, sex, study day (1-7), and treatment group-by-day interaction. The overall estimate for each treatment group were compared; Test type: Superiority; p = 0.0166, Pattern Mixture Model
Statistical Analysis 2: Comparison: DB: Lofexidine HCl 3.2mg Dose vs DB: Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0033, Pattern Mixture Model

2. Secondary Outcome: Completion Status
Description: The percentage of subjects in each treatment arm who receive at least one dose of study medication on Day 7 and complete the 3.5 hour post-dose SOWS-Gossop assessment on Day 7.
Time Frame: Day 7
Population: The percentage of subjects in each treatment arm who complete the double-blind phase of the study (defined as those who receive at least one dose of study medication on Day 7 and complete the 3.5 hour post-dose SOWS-Gossop assessment on Day 7).
Measure: Count of Participants; unit: Participants
Arm/Group | DB: Lofexidine HCl 2.4mg Dose | DB: Lofexidine HCl 3.2mg Dose | DB: Placebo
Number analyzed (Participants) | 229 | 222 | 151
Participants
  Yes/Complete | 95 | 88 | 42
  No/Did Not Complete | 134 | 134 | 109

ADVERSE EVENTS:
Time Frame: Through study completion (14 Days)
Arm/Group | DB: Lofexidine HCl 2.4mg Dose | DB: Lofexidine HCl 3.2mg Dose | DB: Placebo | OL: All Lofexidine HCl
All-Cause Mortality (participants affected / at risk) | 0/229 | 1/222 | 0/151 | 0/83
Serious Adverse Events (participants affected / at risk) | 0/229 | 5/222 | 2/151 | 0/83
Other Adverse Events (participants affected / at risk) | 216/229 | 211/222 | 134/151 | 46/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB: Lofexidine HCl 2.4mg Dose (N=229) | DB: Lofexidine HCl 3.2mg Dose (N=222) | DB: Placebo (N=151) | OL: All Lofexidine HCl (N=83)
Acute hepatitis C (Infections and infestations) | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 2 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB: Lofexidine HCl 2.4mg Dose (N=229) | DB: Lofexidine HCl 3.2mg Dose (N=222) | DB: Placebo (N=151) | OL: All Lofexidine HCl (N=83)
Bradycardia (Cardiac disorders) | 54 | 70 | 8 | 3
Abdominal pain (Gastrointestinal disorders) | 9 | 5 | 9 | 0
Abdominal pain upper (Gastrointestinal disorders) | 19 | 18 | 12 | 4
Diarrhoea (Gastrointestinal disorders) | 51 | 48 | 35 | 5
Dry mouth (Gastrointestinal disorders) | 22 | 24 | 2 | 4
Constipation (Gastrointestinal disorders) | 14 | 17 | 4 | 2
Nausea (Gastrointestinal disorders) | 50 | 27 | 32 | 0
Vomiting (Gastrointestinal disorders) | 23 | 19 | 24 | 1
Pain (General disorders) | 51 | 42 | 36 | 4
Drug withdrawal syndrome (General disorders) | 14 | 14 | 7 | 0
Fatigue (General disorders) | 14 | 16 | 6 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 9 | 9 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 30 | 22 | 25 | 1
Headache (Nervous system disorders) | 30 | 31 | 23 | 4
Sedation (Nervous system disorders) | 29 | 27 | 8 | 1
Dizziness (Nervous system disorders) | 44 | 51 | 4 | 3
Somnolence (Nervous system disorders) | 25 | 29 | 8 | 0
Anxiety (Psychiatric disorders) | 10 | 10 | 10 | 5
Insomnia (Psychiatric disorders) | 117 | 123 | 73 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8 | 6 | 9 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 8 | 4 | 0
Hypertension (Vascular disorders) | 3 | 7 | 15 | 1
Hypotension (Vascular disorders) | 69 | 67 | 2 | 7
Orthostatic hypotension (Vascular disorders) | 67 | 94 | 7 | 4
Tachycardia (Cardiac disorders) | 6 | 2 | 13 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2013-05-06): https://cdn.clinicaltrials.gov/large-docs/86/NCT01863186/Prot_001.pdf
  • Statistical Analysis Plan (2015-01-22): https://cdn.clinicaltrials.gov/large-docs/86/NCT01863186/SAP_000.pdf
  • Informed Consent Form (2013-06-25): https://cdn.clinicaltrials.gov/large-docs/86/NCT01863186/ICF_002.pdf